CLINICAL TRIAL: NCT02767596
Title: A Pilot Single-Arm Open-Label Study to Evaluate the Efficacy of Treatment With Lixisenatide in Diabetes Mellitus Type 2 Patients With Failure of Other GLP-1 Analog
Brief Title: Evaluation of Lixisenatide Efficacy in Diabetes Mellitus Type 2 With Failure of Other GLP-1 Analog
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment rate
Sponsor: Laniado Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIX001
Record Dates: First submitted 2016-04-03; First posted 2016-05-10 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Type 2 Diabetes Mellitus; treatment; GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Insulin Glargine; Insulin Detemir; insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lixisenatide (Experimental): S.C. Lixisenatide 10 mcg for 2 weeks and then 10 mcg for 10 weeks
  Interventions: Drug: Lixisenatide; Drug: Basal insulins

INTERVENTIONS:
Drug: Lixisenatide
  Other Names: Lyxumia
Drug: Basal insulins — patients are on basal insulin treatment
  Other Names: Glargine, Detemir, Degludec

SUMMARY:
The study aims to examine the effectiveness of the short acting GLP-1 analog, Lixisenatide to achieve glycemic control in type 2 diabetes patients, in patients with failure of long acting GLP-1 analog.

Patients who fail to achieve significant improvement in diabetes control on basal insulin and Liraglutide will be switched to basal insulin and lixisenatide treatment for 12 weeks. The primary outcomes will be changes in HBA1C and weight.

ELIGIBILITY:
Inclusion Criteria:

Type Diabetes Mellitus on combination of basal insulin therapy and GLP1 analog, with secondary failure of non-fasting glycemic control

Exclusion Criteria:

* Pregnant or lactating woman
* Renal failure (eGFR<30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c | 16 weeks
Change in body weight | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bildirici Diabetes Center, Laniado Hospital, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No